CLINICAL TRIAL: NCT03487289
Title: Comparison of NOSE and Conventional Methods in Laparoscopic Right Colon Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Ersin Gündoğan, operator doctor, Inonu University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2017/27-5
Record Dates: First submitted 2018-02-03; First posted 2018-04-04 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Surgical Incision
MeSH Terms: conditions — Surgical Wound | interventions — Natural Orifice Endoscopic Surgery; Congresses as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- natural orifice (Experimental): Patients who underwent laparoscopic surgery and removed the specimen from the natural orifice will be gathered. demographic data and perioperative results will be compiled
  Interventions: Procedure: natural orifice
- conventional (No Intervention): patients who underwent laparoscopic surgery and removed specimen with conventional will be gathered. demographic data and perioperative results will be compiled. (conventional extraction is suprapubic or median incision)

INTERVENTIONS:
Procedure: natural orifice — laparoscopic right colon surgery and patients who are removed from the natural orifice and conventional will gather
  Other Names: conventional
  Arms: natural orifice

SUMMARY:
Laparoscopic right hemicolectomy (LRH) is an accepted surgical procedure for several right sided colonic pathologies. Recently the advantages of the intracorporeal ileotransversostomy over the extracorporeal anastomosis is appearing in the literature. Additionally, specimen extraction through the natural orifices is an emerging method when combined with the totally laparoscopic procedures. Our observations on natural orifice surgery was promising . In our daily surgical practice, investigators prefer the intracorporeal anastomosis and this study was conducted to compare the specimen extraction sites after LRH. Here investigators aimed to compare the results of conventional and natural orifice specimen extractions (NOSE) after totally LRHs.

DETAILED DESCRIPTION:
compare the patient-selected NOSE method and conventional method in laparoscopic right colon cancer surgery

ELIGIBILITY:
Inclusion Criteria:

* laparoscopic right hemicolectomy patients

Exclusion Criteria:

* no

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-03-28 (Actual)

PRIMARY OUTCOMES:
VAS control | 6 years
  Visual Analog Score for pain (1-10 score)

CONTACTS AND LOCATIONS:
Overall Officials: Ersin Gündoğan, Principal Investigator — Inonu Unıversity- general surgery
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)